CLINICAL TRIAL: NCT03965260
Title: Data Collection and Identification of Infection-responsible Bacterial Resistances in Cirrhotic Patients
Acronym: RECONNAISSANCE
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: CRC_GHN_2019_005
Record Dates: First submitted 2019-05-23; First posted 2019-05-29 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Cirrhosis
MeSH Terms: conditions — Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Bacteria-infected cirrhotic patients: All kind of etiologies for cirrhosis and all kind of bacterial infections (spontaneous bacterial peritonitis, urinary tract infections, pneumonia, skin and soft tissue infections and spontaneous bacteremia)
  Interventions: Biological: Bacterial samples from blood or peritoneal liquids

INTERVENTIONS:
Biological: Bacterial samples from blood or peritoneal liquids — For each cirrhotic patient hospitalized for a bacterial infection, a blood sample or a peritoneal liquid sample was collected and analyzed for susceptibility, as it is performed in the standard of care. Our department receives only the bacterial results.
  We will then describe the bacterial ecology of the center cirrhotic population in terms of infection acquisition mode, infection site, infection etiology but also drug-resistance.

SUMMARY:
Cirrhotic patients have a high risk of bacterial infection. These infections induce systemic inflammation that can lead to acute liver failure or even acute liver failure associated with multi-visceral failure (Acute-to-Chronic Liver Failure, ACLF) associated with an increased risk of short-term mortality in this population.

The most common infections are spontaneous bacterial peritonitis and urinary tract infections, followed by pneumonia, skin and soft tissue infections and spontaneous bacteremia.

In order to cope with the growing risk of resistant bacterial infections, recommendations from the European Association for the Study of the Liver (EASL) were issued in 2014 and are followed by physicians treating cirrhotic patients. These recommendations advocate taking into account different parameters regarding the best therapeutic strategy to adopt. The site of the infection, the mode of acquisition or the presence or absence of prophylaxis may modify this therapeutic approach to infections of cirrhotic patients to a greater or lesser extent. However, the ecology of a center varies over time, according to the practices of the hospital center and to the different patients in care. It is recommended to update the antibiotic resistance data in order to propose the best therapeutic strategy for these patients.

The study of bacterial resistance in a given care center makes it possible to adapt the recommendations published by EASL in 2014 to the local ecology and to set up protocols of probabilistic antibiotic therapy adapted for a better efficiency.

This descriptive cohort study will determine the local ecology of the center. This will enable the center to assess if the recommended antibacterial strategies correspond to the center bacterial ecology.

DETAILED DESCRIPTION:
Cirrhotic patients have a high risk of bacterial infection. These infections induce systemic inflammation that can lead to acute liver failure or even acute liver failure associated with multi-visceral failure (Acute-to-Chronic Liver Failure, ACLF) associated with an increased risk of short-term mortality in this population.

Cirrhotic patients have a higher risk of infection than the general population because cirrhosis is associated with various changes in the innate and acquired immune response. These changes alter the response to external pathogens, leading to some immunodeficiency (3). Infection is one of the most common risk factors for ACLF and the prevalence of bacterial infections is approximately 25% -46% in hospitalized patients with acute liver decompensation.

The most common infections are spontaneous bacterial peritonitis and urinary tract infections, followed by pneumonia, skin and soft tissue infections and spontaneous bacteremia.

These infections can have various etiologies. The site of infection and the mode of acquisition may affect the risk of infection with resistant bacteria. The increasing diffusion of multidrug-resistant bacteria has made the management of cirrhotic patients and bacterial infections more complex.

Early administration of effective antibiotic therapy is crucial for determining the patient's prognosis. This empirical treatment should be initiated at the earliest after diagnosis of the bacterial infection to avoid an increased mortality risk due to possible septic shock or associated multi-visceral failure (ACLF). The antibiotic treatment administered takes into account the type of infection, the risk of resistant bacterial infection but also the severity of the infection. However, this antibiotic administration can also select multi-resistant bacteria and increase the risk of mortality of the cirrhotic patient.

In order to cope with the growing risk of resistant bacterial infections, recommendations from the European Association for the Study of the Liver (EASL) were issued in 2014 and are followed by physicians treating cirrhotic patients. These recommendations advocate taking into account different parameters regarding the best therapeutic strategy to adopt. The site of the infection, the mode of acquisition or the presence or absence of prophylaxis may modify this therapeutic approach to infections of cirrhotic patients to a greater or lesser extent. However, the ecology of a center varies over time, according to the practices of the hospital center and to the different patients in care. It is recommended to update the antibiotic resistance data in order to propose the best therapeutic strategy for these patients.

The study of bacterial resistance in a given care center makes it possible to adapt the recommendations published by EASL in 2014 to the local ecology and to set up protocols of probabilistic antibiotic therapy adapted for a better efficiency.

This descriptive cohort study will determine the local ecology of the center. This will enable the center to assess if the recommended antibacterial strategies correspond to the center bacterial ecology.

ELIGIBILITY:
Inclusion Criteria:

* Women and men ≥18 years of age
* Cirrhosis diagnosis confirmed with a Doppler and/or a biopsy
* bacterial infection documented with identified germ and susceptibility results
* patient informed and non-opposed to participate

Exclusion Criteria:

* cirrhotic patients with another infection than bacterial infection
* legally protected patients
* patients who expressed their opposition to participate to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Bacteria-infected cirrhotic patients
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Bacterial results | At inclusion
  A cirrhotic patient can have several sampling for bacterial analysis. Blood or peritoneal liquid samples are analyzed to identify the ecology of cirrhotic patients in the center. These bacteria will be described in terms of acquisition mode, infection site and drug-resistance.

CONTACTS AND LOCATIONS:
Locations (1):
- Croix-Rousse Hospital, Hospices Civils de Lyon, Lyon, France

IPD SHARING:
Plan to Share IPD: No